CLINICAL TRIAL: NCT01740687
Title: A Study to Evaluate the Effectiveness of Essure Post-NovaSure Radiofrequency Endometrial Ablation Procedure Following a Successful Essure Confirmation Test
Acronym: ESS-NSPAS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16975
Record Dates: First submitted 2012-11-27; First posted 2012-12-04 (Estimated); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Contraception; Menorrhagia
Keywords: Endometrial Ablation; Permanent Sterilization; Essure; NovaSure; Prevention of Pregnancy
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Essure+NovaSure: The group of women relying on Essure micro-inserts for permanent birth control when NovaSure is performed following a successful Essure Confirmation Test
  Interventions: Device: ESS305 (Essure, BAY1454032); Procedure: NovaSure

INTERVENTIONS:
Device: ESS305 (Essure, BAY1454032) — Essure Permanent Birth Control
Procedure: NovaSure — Nova Sure Endometrial Ablation

SUMMARY:
The purpose of the post approval study is to evaluate the effectiveness and safety of the Essure System when a NovaSure Endometrial Ablation procedure is performed following a successful Essure Confirmation Test.

DETAILED DESCRIPTION:
This study has previously been posted by Conceptus, Inc. After acquiring Conceptus, Inc., Bayer is now the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria from the Essure Permanent Birth Control System Instructions for Use and/or the NovaSure Impedance Controlled Endometrial Ablation (EA) System Instructions for Use and Controller Operator's Manual will apply.
* Women experiencing menorrhagia due to benign causes
* Women who are relying on the Essure micro-inserts for permanent contraception following a successful Essure Confirmation Test (as applicable to the Post Approval Study)
* Women willing to accept the risk of pregnancy while relying on the Essure micro-inserts for prevention of pregnancy following a NovaSure ablation procedure for menorrhagia

Exclusion Criteria:

* All exclusion criteria from the Essure Permanent Birth Control System Instructions for Use and/or the NovaSure Impedance Controlled Endometrial Ablation System Instructions for Use and Controller Operator's Manual will apply.
* Women who previously underwent a fallopian tube sterilization procedure (other than Essure placement)
* Women who present with any other medical complaints, conditions or symptoms unrelated to the Essure System and/or subsequent NovaSure EA including, but not limited to:

  * Gynecological co-morbidities (e.g., pelvic infection, cervicitis, undiagnosed vaginal bleeding, endometrial cancer, myomas, and polyps)
  * Reproductive tract anatomical variants and/or pathology which could make the subject unsuitable for the Essure and/or NovaSure transcervical procedures
* Women currently wearing an intrauterine device and unwilling to have it removed before NovaSure

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Clinics and hospitals
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- United States (17):
  - Aurora, Colorado
  - Ocala, Florida
  - Decatur, Illinois
  - Fort Wayne, Indiana
  - Newburgh, Indiana
  - Easton, Maryland
  - Grand Blanc, Michigan
  - Maplewood, Minnesota
  - Las Vegas, Nevada
  - Neptune City, New Jersey
  - Winston-Salem, North Carolina
  - Englewood, Ohio
  - Mason, Ohio
  - Pottstown, Pennsylvania
  - Nashville, Tennessee
  - Norfolk, Virginia
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 220 participants were screened, of whom 215 participants met all the eligibility criteria at screening. NovaSure procedure was initiated for 211 participants, and 4 participants exited the study before the NovaSure attempt. Two participants for whom the procedure was initiated had the NovaSure procedure terminated before any energy was applied, thus 209 subjects underwent treatment with NovaSure. EA=Endometrial ablation.
Groups:
- Essure + NovaSure: The group of women relying on Essure micro-inserts for permanent birth control when NovaSure was performed following a successful Essure Confirmation Test.
Period: Overall Study
Arm/Group | Essure + NovaSure
Started | 211
Underwent NovaSure EA Treatment | 209
Completed | 174
Not Completed | 37
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 2
Not completed — other reason | 22
Not completed — treatment not received | 2

BASELINE CHARACTERISTICS:
Arm/Group | Essure + NovaSure
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (5.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 207
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 194
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnancies at 1-year Time Point (1-year Pregnancy Rate)
Time Frame: 1 year after NovaSure Endometrial Ablation procedure
Measure: Number; unit: Pregnancy
Arm/Group | Essure + NovaSure
Number analyzed (Participants) | 211
Pregnancy | 0
Statistical Analysis 1: Comparison: Essure + NovaSure; predetermined study success threshold of 2.1% at 1 year; Test type: Other; 95% upper Bayesian credible interval = 1.23 — %

2. Primary Outcome: Number of Pregnancies at 3-year Time Point (3-year Pregnancy Rate)
Time Frame: 3 years after NovaSure Endometrial Ablation procedure
Measure: Number; unit: Pregnancy
Arm/Group | Essure + NovaSure
Number analyzed (Participants) | 211
Pregnancy | 0
Statistical Analysis 1: Comparison: Essure + NovaSure; predetermined study success threshold of 2.8% at 3 years; Test type: Other; 95% upper Bayesian credible interval = 1.33 — %

3. Secondary Outcome: Number of Adverse Events (AEs) When NovaSure Endometrial Ablation Was Performed in the Presence of Essure Inserts
Description: An adverse event (AE) is any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom, or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. A serious adverse event (SAE) is classified as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is another serious or important medical event (IME) as judged by the investigator, or requires intervention to prevent permanent impairment of a body function or damage to a body structure.
Time Frame: After 3-year follow-up
Measure: Number; unit: AEs
Arm/Group | Essure + NovaSure
Number analyzed (Participants) | 211
AEs
  Any AE | 398
  Any SAE | 28

ADVERSE EVENTS:
Time Frame: Up to 3-year follow-up
Arm/Group | Essure + NovaSure
All-Cause Mortality (participants affected / at risk) | 1/211
Serious Adverse Events (participants affected / at risk) | 18/211
Other Adverse Events (participants affected / at risk) | 95/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essure + NovaSure (N=211)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Torsade de pointes (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (3)
Adenomyosis (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essure + NovaSure (N=211)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (5)
Bacterial vaginosis (Infections and infestations) | 3 (4)
Bacterial vulvovaginitis (Infections and infestations) | 4 (4)
Fungal infection (Infections and infestations) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 11 (11)
Vulvovaginal mycotic infection (Infections and infestations) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Migraine (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Stress urinary incontinence (Renal and urinary disorders) | 3 (3)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 3 (4)
Cervical dysplasia (Reproductive system and breast disorders) | 3 (4)
Coital bleeding (Reproductive system and breast disorders) | 4 (4)
Dysmenorrhoea (Reproductive system and breast disorders) | 8 (8)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 7 (8)
Pelvic pain (Reproductive system and breast disorders) | 25 (28)
Uterine haemorrhage (Reproductive system and breast disorders) | 5 (5)
Uterine spasm (Reproductive system and breast disorders) | 6 (6)
Vaginal discharge (Reproductive system and breast disorders) | 15 (17)
Vaginal haemorrhage (Reproductive system and breast disorders) | 10 (10)
Vaginal odour (Reproductive system and breast disorders) | 3 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4)
Hot flush (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT01740687/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT01740687/SAP_001.pdf